CLINICAL TRIAL: NCT05607745
Title: Dietary Counseling Coupled With Fecal Microbiota Transplantation in the Treatment of Obesity and Non-alcoholic Fatty Liver Disease - the DIFTOB Study
Brief Title: Dietary Counseling Coupled With FMT in the Treatment of Obesity and NAFLD - the DIFTOB Study
Acronym: DIFTOB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: Helsinki University Central Hospital (Other); Päijänne Tavastia Central Hospital (Other); University of Helsinki (Other); Kuopio University Hospital (Other); Kuopio Research Institute of Exercise Medicine (Other)
Responsible Party: Principal Investigator, Milla Tauriainen, MD, specialized doctor in gastroenterology and internal medicine, University of Eastern Finland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 13.02.00 1448/2021
Record Dates: First submitted 2022-11-02; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: NAFLD; Fecal Microbiota; Gut Microbiota; Obesity; Dietary Habits; Diet; Fecal Microbiota Transplantation; Glucose Metabolism Disorders; Nutrition, Healthy
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Feeding Behavior; Glucose Metabolism Disorders | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: National multicenter placebo-controlled randomized pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: FMT is given blinded for the participant. The dieticians giving the nutritional advice are also blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT (Active Comparator): Fecal transplantation is given 2:1 compared to placebo transplantation via gastroscopy as a fluid of 100-150ml. Similar healthy diet counseling is given to all participants in both FMT and placebo group.
  Interventions: Other: FMT and placebo
- Placebo (Placebo Comparator): Placebo is brown-colored water and given the same way than fecal transplantation fluid. All study subjects receive similar dietary advice based on healthy diet. Similar healthy diet counseling is given to all participants in both FMT and placebo group.
  Interventions: Other: FMT and placebo

INTERVENTIONS:
Other: FMT and placebo — Similar healthy diet counseling is given to all participants in both FMT and placebo group. FMT to placebo is given in 2:1.

SUMMARY:
There are several studies performed to reveal the linkage between diet, fecal microbiota, and obesity. Human fecal microbiota transplantations in this asset are still scarce. Therefore, this pilot study of FMT from lean to obese people with dietary counseling will increase the knowledge, whether FMT could play a role in the treatment of obesity and NAFLD. Our primary outcome is the changes in glucose metabolism by HOMA-IR.

DETAILED DESCRIPTION:
The prevalence of obesity is rising. In 2015 39% of adults globally, and in 2017 25% of adults in Finland were obese (BMI ≥30kg/m2). Obesity increases the incidence of type 2 diabetes (T2D) and non-alcoholic fatty liver disease (NAFLD).

Obesity associates with decreased gut bacterial diversity, and low microbial gene richness. The diversity of fecal microbiota composition has been shown to alter in human NAFLD. Fecal microbiota transplantation (FMT) from lean vegan donors to those with NAFLD changed fecal microbiota composition and associated with beneficial changes in plasma metabolites in a pilot randomized controlled trial.

Radiological liver imagining for NAFLD is usually performed by ultrasound. Liver elastography evaluates liver stiffness and fibrosis stage. Liver steatosis and fibrosis are known to decrease along weight loss. To our knowledge, only one small study has yet combined FMT and liver imagining in a concept of NAFLD.

Diet influences the gut microbiota. In obesity, the composition of fecal microbiota is altered. Alterations in plasma metabolites derived from gut microbiota and diet have been linked to NAFLD development. The composition of gut microbiome predicts the metabolic response to different dietary interventions in obese individuals.

The key food items of the Healthy Nordic Diet are vegetables, fruit, berries, whole grain products, fish, and rapeseed oil. Abdominal obesity was less abundant in those consuming the Healthy Nordic Diet. Dietary fiber has been associated with metabolically beneficial changes in fecal microbiome. High fat diet has been associated with worsening of fecal microbial composition.

At this moment, the only clinically approved treatment of fecal transplantation (FMT) is recurrent Clostridioides difficile infection. FMT has been studied in asset of obesity and metabolic syndrome in rats, mice and humans. Fecal transplantation from lean donors has been shown to improve insulin sensitivity in obese subjects. Bariatric surgery has been shown to increase fecal microbiota diversity. Giving FMT from bariatric surgery undergone mice or humans lead to weight reduction in the receiver mice. There are studies that have shown no change in glucose metabolism after FMT from lean donor, but also studies with favorable effect on the recipient´s insulin sensitivity and energy expenditure.

The investigators will conduct the randomized controlled one year lasting intervention of dietary advice, where 2:1 participants will be given FMT from lean donor or placebo via gastroscopy to the duodenum. The aim is to investigate the effect of FMT from healthy lean individuals in obese participants receiving dietary counseling.

This study is national multicenter pilot study, where we aim to recruite 54 participants in three different study centers in Kuopio, Lahti and Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥30 kg/m2
* Age 18-75 years
* Signed informed consent
* Ability to take part in a group-based nutrition advice
* Adequate Finnish comprehension (since all advice and materials are in Finnish)

Exclusion Criteria:

* Unable to provide written consent
* Attending another trial or having on-going dietary counseling at the same time
* Pregnancy, breast feeding
* Type I diabetes
* Inflammatory disease
* Liver disease other than NAFLD
* Excess alcohol consumption (more than 20 g/day in females and more than 30 g/day in males, on average)
* Dysmotility of upper GI-tract (e.g. gastroparesis)
* Big hiatal hernia
* History of a severe (anaphylactic) food allergy
* Active, serious medical disease with likely life expectancy less than 5 years
* Severe renal insufficiency (glomerular filtration rate <30%)
* Procedures that have changed the anatomy of GI-tract, including obesity surgery
* Remarkable psychiatric disorders, dementia and other diseases or conditions that could affect to the study subject´s compliance to the study
* Systemic antibacterial treatments

  * three months before the study or during the study
  * chronic or recurrent bacterial infection for which antimicrobial medications are repeatedly used
* Contraindication for gastroscopy
* Central anesthesia needed for gastroscopy
* Medications for losing weight (bupropion/naltrexon, orlistat, liraglutide)
* Intention to obesity surgery.

Eligibility is evaluated by a doctor in each research unit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
A change in HOMA-IR | at week 12 and at week 52
  A change in HOMA-IR at week 12 and week 52 in both study groups and hypothetically more in those with FMT compared to those with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Milla-Maria Tauriainen, MD, Principal Investigator — Kuopio University Hospital
Locations (3):
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - University of Eastern Finland, Kuopio
  - Lahti Central Hospital, Lahti

IPD SHARING:
Plan to Share IPD: No
RedCap will be used across different research sites.